CLINICAL TRIAL: NCT03261973
Title: Esophageal Deviation in Atrial Fibrillation Ablation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Moussa C Mansour, Principal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2017P001544
Record Dates: First submitted 2017-08-21; First posted 2017-08-25 (Actual); Results first posted 2021-06-30 (Actual); Last update posted 2021-06-30 (Actual); Status verified 2021-06

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- DV8 esophageal deviation tool (Other): This is a non-randomized one arm study.
  Interventions: Device: DV8

INTERVENTIONS:
Device: DV8 — DV8 esophageal deviation tool

SUMMARY:
Catheter ablation with pulmonary vein (PV) isolation is a commonly performed strategy employed for the treatment of atrial fibrillation (AF). However, ablation in the posterior wall of the left atrium can cause thermal injury to the esophagus. Thermal injury is very common and occurs in up to 40% of AF ablations per some studies. When significant thermal injury to the esophagus occurs, two significant complications can arise: 1) the formation of an atrio-esophageal fistula, and 2) gastrointestinal dysmotility. While the occurrence of fistula is rare, it is a very important complication since it is often fatal. Currently luminal esophageal temperature monitoring is the most commonly employed modality to prevent such injury. However, there are limitations to its use, and atrio-esophageal fistulas continue to be a major problem in AF ablation even when using esophageal temperature monitoring. Esophageal deviation using either a Transesophageal echocardiogram (TEE) or Esophagogastroduodenoscopy (EGD) probe has been described in the literature, but the effectiveness and practicality of these techniques are suboptimal, and have therefore precluded their use in routine clinical practice. Recently, esophageal deviation using off-the-shelf equipment (a soft thoracic tube and endotracheal stylet) was tested in the randomized double-blind multicenter study "Deviating the Esophagus in Atrial Fibrillation Ablation (DEVIATE-AF)". In that study the standard practice (i.e., use of luminal esophageal temperature monitoring) was compared to esophageal deviation using off-the-shelf equipment. The results were very encouraging showing that esophageal deviation allowed for significant reductions in esophageal temperature and proportion of premature ablation terminations. Importantly, esophageal deviation allowed the isolation all PVs in the treatment group, which was not the case in the control group. One major limitation in the DEVIATE-AF trial was that off-the-shelf equipment tool was challenging to use. The aim of the Esophageal Deviation in Atrial Fibrillation Ablation study is to test the feasibility and safety of moving the esophagus using a specialized esophageal deviation tool (DV8, Manual Surgical Sciences, Minneapolis, MN).

ELIGIBILITY:
INCLUSION CRITERIA

* A maximum of up to 54 patients will be enrolled in this prospective single-center single-arm study. Patients undergoing AF ablation (including paroxysmal and persistent AF) will be included in this study. Consistent with the current definitions, paroxysmal AF are episodes that will self-terminate in less than 24 hours. Persistent AF, is defined as ≥1 documented AF lasting >1week in duration or lasting less than 7 days but requiring electrical or pharmacological cardioversion to sinus rhythm.
* Age >18 - Age < 80 yr
* Documentation of atrial fibrillation (AF)
* General anesthesia
* All patients must understand and adhere to the requirements of the study and be willing to comply with the post study follow-up requirements.

EXCLUSION CRITERIA

* Any reversible cause of AF (post-surgery, thyroid disorder, etc.)
* INR (international normalized ratio) > 4.0 at the time of the procedure
* History of (H/o) of severe esophageal ulcers, strictures, varices, bleeding, laceration or perforation, esophagitis
* Severe Gastroesophageal Reflux Disease (GERD)
* H/o esophageal surgery or any esophageal banding or cautery
* H/o chest radiation
* Significant abnormality on Swallowing Impairment Score
* Mental impairment precluding signing consent or completing follow up
* Patients with any other significant uncontrolled or unstable medical condition
* Women who are known to be pregnant or have had a positive β-HCG (Human Chorionic Gonadotropin) test within 7 days prior to procedure
* Presence of left atrial thrombus

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2017-11-17 (Actual); Primary Completion 2020-06-15 (Actual); Study Completion 2020-06-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- DV8 Esophageal Deviation Tool: This is a non-randomized one arm study.
  Arm: usage of the DV8 esophageal deviation tool during the ablation procedure
Period: Overall Study
Arm/Group | DV8 Esophageal Deviation Tool
Started | 47
Completed | 43
Not Completed | 4

BASELINE CHARACTERISTICS:
Arm/Group | DV8 Esophageal Deviation Tool
Number analyzed (Participants) | 43
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.9 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 31
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Minimum Distance of 1 cm Esophageal Deviation Between the Ablation Line for the Ipsilateral Pulmonary Vein (PV) Pairs and the Trailing Edge of the Esophagus.
Time Frame: during Atrial Fibrillation (AF) ablation procedure (intraoperative)
Measure: Count of Participants; unit: Participants
Arm/Group | DV8 Esophageal Deviation Tool
Number analyzed (Participants) | 43
Participants | 42

2. Secondary Outcome: Number of Participants With an Average Distance of 2 cm Esophageal Deviation From the Ablation Line for the Ipsilateral PV Pairs.
Time Frame: during AF ablation procedure
Measure: Count of Participants; unit: Participants
Arm/Group | DV8 Esophageal Deviation Tool
Number analyzed (Participants) | 43
Participants | 9

3. Secondary Outcome: Number of Participants Who Experienced Esophageal Laceration
Time Frame: within 1-90 days of the procedure
Measure: Count of Participants; unit: Participants
Arm/Group | DV8 Esophageal Deviation Tool
Number analyzed (Participants) | 43
Participants | 0

4. Secondary Outcome: Number of Participants With PV Reconnection Assessed by Adenosine Infusion
Time Frame: during AF ablation procedure
Measure: Count of Participants; unit: Participants
Arm/Group | DV8 Esophageal Deviation Tool
Number analyzed (Participants) | 43
Participants | 10

5. Secondary Outcome: Fluoroscopy Time Measured for the Whole Procedure
Time Frame: during AF ablation procedure
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | DV8 Esophageal Deviation Tool
Number analyzed (Participants) | 43
minutes | 23.8 (8.1)

6. Secondary Outcome: Procedure Duration Measured From the Initial Groin Stick to Catheter Removal
Time Frame: during the AF ablation procedure
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | DV8 Esophageal Deviation Tool
Number analyzed (Participants) | 43
minutes | 212 (32)

7. Secondary Outcome: Ablation Time Assessed by the Total Duration of Radiofrequency Energy Delivery
Time Frame: during the AF ablation procedure
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | DV8 Esophageal Deviation Tool
Number analyzed (Participants) | 43
minutes | 53.2 (16.2)

ADVERSE EVENTS:
Time Frame: The duration of the study was 3 months
Arm/Group | DV8 Esophageal Deviation Tool
All-Cause Mortality (participants affected / at risk) | 0/43
Serious Adverse Events (participants affected / at risk) | 0/43
Other Adverse Events (participants affected / at risk) | 2/43
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | DV8 Esophageal Deviation Tool (N=43)
Gastroparesis (Gastrointestinal disorders) | 1
Pericarditis (Cardiac disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-07-18): https://cdn.clinicaltrials.gov/large-docs/73/NCT03261973/Prot_SAP_000.pdf